CLINICAL TRIAL: NCT03915353
Title: Evaluation Of Vestibular Functions and Balance in Edirne Band Musicians
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Halit SELÇUK, Research Assisstant, Trakya University
Other Study IDs: 2017/234
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Vestibular Disorder
Keywords: Noise; Balance; Quality of Life
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment: No interventions
  Interventions: Other: No Intervention
- Control: No interventions
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
It has been stated that intense noise may affect the peripheral vestibular system and consequently cause problems in balance mechanisms. The aim of this study was to investigate the effects of exposure to chronic noise on vestibular functions and balance in Edirne Band musicians.

Twenty-two individuals working in the Edirne Band for at least 5 years and over 18 years of age and a control group of 22 individuals working at Trakya University and with similar sociodemographic characteristics to the experimental group were included. The socio-demographic questionnaire was used to inquire about the demographic characteristics of individuals and alcohol-cigarette use, the Activity-Specific Balance Confidence Scale to assess how they felt about the balance, and the Dizziness Handicap Inventory to determine the quality of life-related to dizziness. A 3D ultrasonic system was used to assess the static and dynamic balance of the individuals.

DETAILED DESCRIPTION:
Chronic exposure to intense noise causes temporary or permanent hearing loss. The effects of exposure to intense noise on the auditory system are well explained, but the number of studies that observes the effects of noise on the vestibular system is limited. It has been stated that intense noise may affect the peripheral vestibular system and consequently cause problems in balance mechanisms. The aim of this study was to investigate the effects of exposure to chronic noise on vestibular functions and balance in Edirne Band musicians.

Twenty-two individuals working in the Edirne Band for at least 5 years and over 18 years of age who did not have a diagnosed vestibular disorder, no cervical vertebrae problem, no musculoskeletal system problems during the evaluation and a control group of 22 individuals working at Trakya University and with similar sociodemographic characteristics to the experimental group were included in the study. The socio-demographic questionnaire was used to inquire about the demographic characteristics of individuals and alcohol-cigarette use, the Activity-Specific Balance Confidence Scale to assess how they felt about the balance, and the Dizziness Handicap Inventory to determine the quality of life-related to dizziness. A 3D ultrasonic system was used to assess the static and dynamic balance of the individuals.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Had at least for 5 years of experience at the Edirne Band
* Volunteering to participate in the study

Exclusion Criteria:

* Diagnosed vestibular disease
* Cervical spine problems during the evaluation
* Musculoskeletal problems during the evaluation

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: 22 males working as a musician in Edirne Band and a control group working in Trakya University with similar sociodemographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Romberg Test | 20 minutes after obtaining socio-demographic information, participants who met the inclusion criteria included in the test.
  Romberg test was assessed in the Zebris system. All measurements were performed in a quiet environment. For the Romberg test, the patient was asked to stay still for 60 seconds with his eyes closed, his feet contiguous, and his shoulders at 90 degrees flexion.
Unterberger's Test | 25 minutes after obtaining socio-demographic information, participants who met the inclusion criteria included in the test.
  Unterberger's test was assessed in the Zebris system. All measurements were performed in a quiet environment. For the Unterberger's test, subjects closed their eyes and began stepping in place for 60 seconds with shoulder at 90 degrees flexion, arms extended forward

SECONDARY OUTCOMES:
Activities-Specific Balance Confidence Scale | 5 minutes after obtaining socio-demographic information.
  ABC developed by Myers and Powel is a questionnaire based on evaluations of how confidently they can do 16 activities within and outside the house. Each activity scored between 0 (insecure) and 100 (completely confident). The total score (0-1600) is divided into 16 and the individual's ABC score is obtained. It has been shown to be reliable in patients with vestibular dysfunction. Higher values in ABC Scale represent a better outcome.
Dizziness Handicap Inventory | 10 minutes after obtaining socio-demographic information.
  DHI is a questionnaire that evaluates the quality of life and the disability caused by complaints related to dizziness and imbalance. DHI, developed by Jacobson and Newman, is a 25-item scale that identifies sensory and functional outcomes in patients with vestibular system problems, as well as factors affecting dizziness and balance disorder. Three subscales are aimed to determine the physical, sensory and functional effects of vestibular system diseases. The subscale scores which are considered as the limit for the determination of disability are 28 points for physical disability and 36 points for functional and sensory disability. Higher scores indicate that the person has more disability due to dizziness. According to the total score taken from the scale, people have divided into 3 groups; 0-30 points (mild disability), 31-60 points (moderate disability), 61-100 points (severe disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No